CLINICAL TRIAL: NCT03201562
Title: A Single-Center, Double-Masked Evaluation of the Efficacy and Safety of PRX-100 in the Treatment of Early to Moderate Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRX100.FDAIIb
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — aceclidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aceclidine+tropicamide combination (Experimental): Aceclidine+tropicamide combination single dose (PRX-100 Ophthalmic Solution)
  Interventions: Drug: Aceclidine+tropicamide combination
- Aceclidine (Active Comparator): Aceclidine single dose
  Interventions: Drug: Aceclidine
- Vehicle (Sham Comparator): Vehicle single dose
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Aceclidine+tropicamide combination — Ophthalmic Solution
  Other Names: PRX-100
  Arms: Aceclidine+tropicamide combination
Drug: Aceclidine — Ophthalmic Solution
  Arms: Aceclidine
Drug: Vehicle — Ophthalmic Solution
  Arms: Vehicle

SUMMARY:
To evaluate the safety and efficacy of PRX-100 compared with aceclidine alone and vehicle in the treatment of early to moderate presbyopia.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent and sign Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed;
2. Be able and willing to follow all instructions and attend study visits;
3. Be 48-64 years of age of either sex and any race or ethnicity at visit 1;
4. Be an early to moderate presbyope determined by screening monocular best-corrected distance visual acuity (VA) at 45 cm
5. Be able and willing to avoid all disallowed medications for the appropriate washout period and during the study without significant risk to the subject.

Exclusion Criteria:

1. Be a female of childbearing potential who is currently pregnant, nursing or planning a pregnancy;
2. Have known contraindications or sensitivity to the use of any of the study medications(s) or their components;
3. Have an active ocular infection at visit 1 (bacterial, viral or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation (eg, moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis, scleritis, uveitis) in either eye;
4. Have moderate or severe dry eye;
5. Have clinically significant abnormal lens findings (eg cataract) including early lens changes and/or any evidence of a media opacity in either eye;
6. Have dark-adapted pupillometry measurements of < 4.0 mm in either eye;
7. Have intraocular pressure (IOP) that is less than 5 millimeters of mercury (mmHg) or greater than 22 mmHg in either eye documented at visit 1, or have a prior diagnosis of ocular hypertension or glaucoma or currently being treated with any type of topical IOP lowering (glaucoma) medication at visit 1;
8. Have abnormal findings on dilated fundus exam in either eye documented within 3 months of visit 1 or a known history of retinal detachment or clinically significant retinal disease in either eye;
9. Have a known history or diagnosis in the past of: iritis, scleritis or uveitis, whether active or inactive;
10. Have had surgical intervention (ocular or systemic) within 6 months prior to visit 1, or planned surgical intervention within 30 days after visit 4;
11. Have undergone refractive eye surgery (incisional keratotomy, photorefractive keratectomy [PRK], laser in situ keratomileusis [LASIK], laser-assisted sub-epithelial keratectomy [LASEK]), corneal inlay procedures, cataract extraction, or intraocular lens placement;
12. Use artificial tears or lubricant eye ointment on a daily basis;
13. Have an inability or refuse to discontinue soft contact lens wear 7 days prior to study visit 1 and rigid gas permeable (RGP) contact lens wear 14 days prior to visit 1 and during the study;
14. Use any of the following disallowed medications during the 2 weeks (14 days) prior to visit 1 and during the study:

    1. narcotic (opiate class) pain medication (eg, codeine, OxyContin®, Vicodin®, Tramadol®)
    2. bladder medication (eg Urecholine®, bethanechol)
    3. antipsychotics
    4. antidepressants
    5. attention -deficit/hyperactivity disorder (ADHD) medications
    6. alpha-blockers (eg, tamsulosin, Flomax®, Jayln®, Uroxatral®, Rapaflo®)
    7. anticholinergics (eg, atropine, belladonna, benztropine, dicyclomine, donepezil, hyoscyamine, propantheline, scopolamine, trihexphenidyl)
    8. muscarinic receptor agonists or cholinergic agonists (eg, Salagen®, Evoxac®)
    9. over-the-counter (OTC) or prescription antihistamines or decongestants
    10. any prescribed topical ophthalmic medications
    11. recreational drug use (eg, marijuana, methadone, heroin, cocaine);
15. Have a diagnosis of diabetes mellitus or a history of elevated blood sugar;
16. Have a condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation, including but not limited to unstable: cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 48 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crossover Sequence 1: Aceclidine+tropicamide combination Visit 1, Aceclidine Visit 2, Vehicle Visit 3
- Crossover Sequence 2: Aceclidine Visit 1, Vehicle Visit 2, Aceclidine+tropicamide combination Visit 3
- Crossover Sequence 3: Vehicle Visit 1, Aceclidine+tropicamide combination Visit 2, Aceclidine Visit 3
Period: Overall Study
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3
Started | 18 | 20 | 20
Completed | 18 | 19 | 16
Not Completed | 0 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Sequence 1 | Crossover Sequence 2 | Crossover Sequence 3 | Total
Number analyzed (Participants) | 18 | 20 | 20 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (3.29) | 55.7 (4.28) | 56.2 (4.51) | 55.6 (4.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 11 | 27
  Male | 9 | 13 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 16 | 20 | 20 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 15 | 18 | 20 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With at Least a 3 Line (15 Letter) Improvement in Near Visual Acuity in the Study Eye
Description: Proportion of subjects with at least a 3 line (15 letter) improvement in near visual acuity in the study eye at 1 hour post-treatment in the mITT population
Time Frame: 1 hour post-treatment
Population: The treatment crossover design allowed for each treatment to be analyzed in all 58 subjects. The primary efficacy analysis was performed on a mITT population of subjects meeting the baseline criteria.
Measure: Number; unit: percentage of participants
Groups:
- Aceclidine+Tropicamide Combination: Aceclidine+tropicamide combination single dose
Arm/Group | Aceclidine+Tropicamide Combination | Aceclidine | Vehicle
Number analyzed (Participants) | 36 | 36 | 42
percentage of participants | 47.22 | 47.22 | 2.38
Statistical Analysis 1: Comparison: Aceclidine+Tropicamide Combination vs Vehicle; Test type: Superiority; p = 0.0009, Generalized Estimating Equation (GEE); GEE model includes 3-line improvement as response variable with sequence, period, treatment as fixed effect, subject within sequence as random effect; Odds Ratio (OR) = 38.436, 90% CI 2-sided [6.262 to 235.936]
Statistical Analysis 2: Comparison: Aceclidine vs Vehicle; Test type: Superiority; p = 0.0012, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 36.893, 90% CI 2-sided [5.936 to 229.310]
Statistical Analysis 3: Comparison: Aceclidine+Tropicamide Combination vs Aceclidine; Test type: Superiority; p = 0.9298, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.042, 90% CI 2-sided [0.485 to 2.239]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 50 days.
Description: Safety population includes all randomized subjects who receive at least one dose of the study medication.
Arm/Group | Aceclidine+Tropicamide Combination | Aceclidine | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 22/54 | 22/54 | 10/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aceclidine+Tropicamide Combination (N=54) | Aceclidine (N=54) | Vehicle (N=57)
Instillation site pain (mild) (Eye disorders) | 17 | 16 | 6
Instillation site pain (moderate) (Eye disorders) | 2 | 5 | 4
Ocular hyperaemia (Eye disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must not present the study results until the aggregate multi-site study results are published. The PI must submit to sponsor any proposed publication or presentation at least 60 days prior to the submission. Sponsor may require the delay of publication or presentation for an additional period of time not to exceed 120 days for the purposes of filing patent applications to patentable subject matter or the resolution of any inaccuracies or misleading statements.

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03201562/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03201562/SAP_001.pdf